CLINICAL TRIAL: NCT02449564
Title: The Pilot Study Evaluate the Safety and Efficacy of Sirolimus in Patients With PIK3CA Mutation and/or PIK3CA Amplification Refractory Solid Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, MD,PhD, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-10-030
Record Dates: First submitted 2015-05-14; First posted 2015-05-20 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sirolimus (Experimental): sirolimus 1mg daily
  Interventions: Drug: sirolimus

INTERVENTIONS:
Drug: sirolimus — sirolimus 1mg daily

SUMMARY:
This study is a single-arm, phase II study of sirolimus in patient with PIK3CA mutation and PIK3CA amplication Refractory solid tumors.

sirolimus 1mg will be administered orally qd daily.

To investigate the efficacy of sirolimus in patients with PIK3CA mutation and PIK3CA amplication Refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of fully informed consent prior to any study specific procedures.
2. Patients must be ≥20 years of age.
3. PIK3CA amplification and/or PIK3CA mutation Refractory Solid Tumors.
4. ECOG performance status 0-2.
5. Have measurable or evaluated disease based on RECIST1.1. as determined by investigator.
6. Adequate Organ Function Laboratory Values

   * Absolute neutrophil count ≥ 1.5 x 109/L, Hemoglobin ≥ 9g/dL, Platelets ≥ 100 x 109/L
   * bilirubin ≤ 1.5 x upper limit of normal AST/ALT ≤ 2.5 x upper limit of normal (5.0 X upper limit of normal , for subjects with liver metastases)
   * creatinine ≤1.5 x UNL
7. Patients of child-bearing potential should be using adequate contraceptive measures (two forms of highly reliable methods) should not be breast feeding and must have a negative pregnancy test prior to start of dosing.
8. Adequate heart function.

Exclusion Criteria:

1. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≤5 years.
2. Has known active central nervous system (CNS) metastases.
3. Has an active infection requiring systemic therapy.
4. Pregnancy or breast feeding
5. Patients with cardiac problem.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-11-24 (Actual); Primary Completion 2017-09-27 (Actual); Study Completion 2017-11-03 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 24 weeks

SECONDARY OUTCOMES:
overall response rate | 24 weeks
overall survival | 24 weeks
Time to progressive | 24 weeks
Number of subjects with Adverse Events as a measure of toxicity profile | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jee yun Lee, MD,Ph.D., Principal Investigator — Samsung Medical Center,Seoul,Korea
Locations (1):
- Samsung Medical center, Seoul, South Korea